CLINICAL TRIAL: NCT03927495
Title: Phase II Study of KN046 in Patients With Recurrent or Metastatic Esophageal Squamous Cell Carcinoma to Evaluate Safety, Efficacy and Tolerance
Brief Title: KN046 in Patients With Recurrent or Metastatic Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: First Affiliated Hospital of Suzhou Medical College (Other)
Responsible Party: Principal Investigator, Xiaolong Fu, Director, Department of Radiation Oncology, Shanghai Chest Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KN046-IST-01
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — TP protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concurrent chemoradiotherapy and KN046 (Experimental): Participants in the Arm I will receive chemoradiotherapy and concurrent KN046. Radiotherapy will be completed within the four-cycle of chemotherapy.
  Interventions: Drug: KN046; Radiation: palliative radiotherapy
- chemoradiotherapy and sequential KN046 (Experimental): Participants in the Arm II will receive chemoradiotherapy and sequential KN046. Radiotherapy will be completed within the four-cycle of chemotherapy.
  Interventions: Radiation: palliative radiotherapy; Drug: KN046

INTERVENTIONS:
Drug: KN046 — Cisplatin+paclitaxel will be administered once every three weeks for four cycles. During the period of radiotherapy, KN046 will be administered once every two weeks until progressive disease, unacceptable toxicity or up to 2 years.
  Other Names: Cisplatin+paclitaxel
  Arms: Concurrent chemoradiotherapy and KN046
Radiation: palliative radiotherapy — 3D conformal radiation therapy will be administered for esophageal lesion or nearby lymph node. Stereotactic body radiation will be administered for metastatic lesion.
Drug: KN046 — Cisplatin+paclitaxel will be administered once every three weeks for four cycles. After completion of radiotherapy, KN046 will be administered once every two weeks until progressive disease, unacceptable toxicity or up to 2 years.
  Other Names: Cisplatin+paclitaxel
  Arms: chemoradiotherapy and sequential KN046

SUMMARY:
This is an open-label, phase II study of KN046 combined with chemotherapy and palliative radiotherapy in patients with recurrent or metastatic esophageal squamous cell carcinoma to evaluate the safety, efficacy and tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Signed inform consent form(ICF)
* Age ≥ 18 years and ≤ 75 years, male or female
* Histologically or cytologically documented recurrent or metastatic esophageal squamous cell carcinoma, with indications of radiotherapy and without prior systemic treatment
* At least one measurable lesion according to Response Evaluation Criteria In Solid Tumors（RECISIT） v 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ function
* Female patients and males with partners of childbearing potential should be using highly effective contraceptive measures (failure rate of less than 1% per year). Contraception should be continued for a period of 24 weeks after dosing has been completed.
* Ability to comply with treatment, procedures and pharmacokinetics (PK) sample collection and the required study follow-up procedures

Exclusion Criteria:

* Known brain metastasis or another Central Nervous System (CNS) metastasis that is either symptomatic or untreated.
* Patients who are participating or have participated in a study of an investigational drug within 4 weeks prior to the first dose of trial treatment.
* Patients who have received immune checkpoint proteins/antibody/medicine for treatment.
* Patients who have interstitial lung disease, or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management.
* Subjects with active autoimmune diseases or history of autoimmune diseases should be excluded
* Active Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) infection.
* Known HIV infection or known history of acquired immune deficient syndrome (AIDS)
* Any unresolved the Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥ 2 toxicities from prior anti-cancer therapy except for vitiligo, alopecia
* Patients who have serious hypersensitive reaction to monoclonal antibodies and have history of uncontrolled allergic asthma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-22 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
dose-limiting toxicity KN046 | 28 days after first dose
6-month progression free survival rate assessed by investigator based on RECIST 1.1 | 6 months after first dose
Objective response rate assessed by investigator based on RECIST 1.1 | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Suzhou University, Suzhou, China